CLINICAL TRIAL: NCT02554526
Title: Basic Study on Novel Therapeutic Strategy With Bypassing Agent Therapy in Hemophilia A Patients With Inhibitors
Brief Title: Basic Study of Combination Therapy Based on APCC-induced FVllI Activation in Hemophilia A Patients With Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nara Medical University (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Keiji Nogami, MD,PhD, Associate Professor, Nara Medical University
Other Study IDs: J150100036
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Hemophilia A With Inhibitor
Keywords: hemophilia A; inhibitor; bypassing therapy; factor VIII
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Combination therapy: Effects of aPCC reaction in the presence of FVIII

SUMMARY:
Using whole blood samples and plasma samples obtained from some hemophilia A patients with inhibitors, the investigators will perform the coagulation assessment in the co-presence of aPCC and factor VIII by comprehensive coagulation assays and flow chamber analysis under blood flow conditions.

DETAILED DESCRIPTION:
Comprehensive coagulation assays using recently popular rotational thromboelastometry (ROTEM), factor Xa/thrombin/plasmin generation test, and coagulation wave analysis and recently developed flow chamber system under blood flow conditions (T-TAS®) will be used. A bypassing agent, aPCC (Feiba®) and recombinant factor VIII (Advate®) will be added ex vivo to whole blood and plasma samples from patients with hemophilia A with inhibitors to compare with the coagulation effects of aPCC in the presence of factor VIII and those of aPCC in its absence under the conditions close to the physiological condition. Furthermore, the difference in the coagulation effects by the difference in inhibitor epitopes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A with inhibitors (Inhibitor titer; >0.5 Bethesda U/ml)
* Patients with agreement consents with the patients signatures

Exclusion Criteria:

* Patients that do not fill the conditions described above

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We guess that there are approximately 200-300 hemophilia A patients with inhibitors in our country. We have approximately 20 out-patients in our hospital. Based on this information, we set up the patients subjects (n=10).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of coagulation effects using patients' plasmas by FXa/thrombin/plasmin generation tests and clot waveform analysis | up to 10 months
Evaluation of coagulation effects using patients' whole bloods by ROTEM and T-TAS | up to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Midori Shima, MD, PhD, Study Director — Nara Medical University
Locations (1):
- Department of Pediatrics, Kashihara, Nara, Japan